CLINICAL TRIAL: NCT06699771
Title: A Phase 1, Multicenter Trial to Assess the Safety, Tolerability, and Preliminary Efficacy of GCC2005 With Lymphodepleting Chemotherapy in Treatment of Patients With Relapsed or Refractory NK and T-cell Malignancies
Brief Title: Phase 1 to Investigate the Safety, Tolerability, and Efficacy of GCC2005 in Patients With R/R NK and T-cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GC Cell Corporation (Industry)
Collaborators: Artiva Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCC2005A-P101
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-10

CONDITIONS: Lymphoma, T-Cell
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: The dose-escalation part of the study (Phase 1a) employs a 3+3 design to determine the DLT of GCC2005.
  The dose-expansion part of the study (Phase 1b) will enroll patients in two cohorts to determine MTD and RP2D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase 1a Dose Escalation and Phase 1b Dose Expansion (Experimental): Dose Confirmation of GCC2005 in Relapsed or Refractory NK and T-cell Malignancies
  Interventions: Drug: GCC2005; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: GCC2005 — CAR-NK Cell Therapy
Drug: Cyclophosphamide — Lymphodepleting chemotherapy
Drug: Fludarabine — Lymphodepleting chemotherapy

SUMMARY:
This is a Phase 1 (a and b), first in human (FIH), single-arm, open-label, multicenter study to evaluate the safety, tolerability and efficacy of GCC2005 in the treatment of patients with relapsed/refractory (R/R) NK or T-cell malignancies who have received at least two prior lines of therapy.

DETAILED DESCRIPTION:
The purpose of the study is to assess the safety, tolerability, and preliminary efficacy of GCC2005 in treatment of patients with relapsed or refractory NK cell and T-cell malignancies expressing CD5. Phase 1a of the study will be conducted to establish a dose range that is well tolerated by the majority of patients and to provide a safety profile of GCC2005 in target patient population. Phase 1b of the study is planned to conduct dose optimization to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory CD5+ NK and T-cell originated malignancies (per WHO classification 2017).
* Patients with relapsed or refractory disease previously treated with two or more lines of standard chemotherapies and there is no longer any treatment option considered as assessed by the Investigator.
* According to the Lugano classification, patients having lesion/nodules ≥ 1 with diameter longer than 1.5 cm for nodal lesions and longer than 1.0 cm for extranodal lesions, and the boundaries are clearly shown.
* Patient has a performance status of 0, 1, or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
* Patients who satisfy the criteria defined in the protocol.
* Contraceptive use by men and women must be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Has T-ALL/T-LBL or CTCL.
* Patient with CNS lymphoma or any involvement of the CNS.
* Patient who had a prior history of another malignancy over the last 3 years.
* Patients who have used hematopoietic growth factor therapy within 14 days prior to Screening.
* Patients who have had prior CAR-T or CAR-NK therapies.
* Presence of uncontrolled fungal, bacterial, viral infection or other infection requiring IV antimicrobials for management
* Patients with previous allogenic organ transplantation
* Patients with previous diagnosis of primary immunodeficiency or currently undergoing therapy of primary immunodeficiency.
* Patients with acute GvHD ≥ Grade 3 or extensive chronic GvHD within 2 weeks of lymphodepletion.
* Patients with known active Hepatitis B or C
* Patients with presence of Grade 2 or greater toxicity from the previous treatment.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Safety: Frequency, severity, and persistence of AEs and AEs Grade 3 or higher | From the time of enrollment through End of Study (up to 18 months per patient)
  To evaluate the safety and tolerability of GCC2005 in patients with relapsed/refractory NK/T cell malignancies.
  Frequency, severity, and persistence of AEs and AEs Grade 3 or higher using NCI CTCAE ver5.0 including CRS, and neurotoxicity based on the ASTCT criteria and acute GvHD based on the Mount Sinai Acute GvHD MAGIC guidance and chronic GvHD based on the National Institutes of Health 2014 criteria, incidence of TEAEs.
  Dose-limiting toxicities (DLTs)
To determine MTD and RP2D: Safety(based on frequency, severity, and persistence of AEs and AEs Grade 3 or higher), efficacy (based on ORR) and pharmacokinetics | From the time of enrollment through End of Study (up to 18 months per patient)
  To determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D)
  Frequency, severity, and persistence of AEs and AEs Grade 3 or higher using NCI CTCAE ver5.0 including CRS, and neurotoxicity based on the ASTCT criteria and acute GvHD based on the Mount Sinai Acute GvHD MAGIC guidance and chronic GvHD based on the National Institutes of Health 2014 criteria, incidence of TEAEs.
  Dose-limiting toxicities (DLTs)

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Seoul National University Hosptial, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No